CLINICAL TRIAL: NCT03137043
Title: Observational Study to Describe the Prevalence of Severe Asthma in Spanish Hospitals
Brief Title: Prevalence of Severe Asthma in Spanish Hospitals
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Quintiles IMS (Unknown)
Responsible Party: Sponsor
Other Study IDs: 205807
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Asthma
Keywords: GINA guidelines; Prevalence; Mepolizumab; severe asthma; Spain
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Asthmatic Subjects: Subjects requiring high dose inhaled corticosteroids (ICS) plus a second controller (and/or systemic glucocorticosteroids) to prevent it from becoming 'uncontrolled' or which remains 'uncontrolled' despite the therapy.
  Interventions: Other: Questionnaire; Other: Software of Big Data
- Non-Severe Asthmatic Subjects: Subjects with intermittent, persistent mild or moderate asthma.
  Interventions: Other: Questionnaire; Other: Software of Big Data

INTERVENTIONS:
Other: Questionnaire — Subjects will be given an Electronic Case Report Form (eCRF) with a series of questionnaire such as Asthma Control Test, Morisky-Green Questionnaire and St George's Respiratory Questionnaire.
Other: Software of Big Data — Software of big data is a powerful data treatment algorithm works closely with Spanish Data Protection Agency as an example on how to reuse clinical information without conflicting with necessary data privacy. The system will process a vast amount of information (big data), so that the impact of random errors will be minimized.

SUMMARY:
Asthma is a chronic disease. Prevalence of asthma in 2014 among Spanish population was 5%, of which 10% were diagnosed with severe asthma. According to Spanish National Guideline for the Management of Asthma (GEMA) 4.1 criteria, asthma can be classified according to its severity (intermittent, mild persistent, moderate persistent or severe persistent) or level of asthma control (controlled, partly controlled or uncontrolled). This Guideline describes that only 1 in 10 subjects with severe asthma is well controlled, meaning that there is a 90% prevalence of non-controlled severe asthma.

This prospective, non-interventional, observational, multicenter and case-control study aims to assess the prevalence of severe asthma in Spanish Hospitals. The study will describe the characteristics of severe versus non-severe asthmatic subjects, assess their eligibility to receive biological treatments approved for this disease, resource consumption and evaluate the most prevalent phenotypes of severe asthma in Spain. Enrolled subjects will be divided into two cohorts, based on asthma severity according to the Global Initiative for Asthma (GINA) and the International European Respiratory Society (ERS)/American Thoracic Society (ATS) Guidelines. Cohort A: subjects diagnosed of severe asthma and Cohort B: subjects with non-severe asthma. Approximately 320 severe asthmatic subjects and 160 non-severe asthmatic subjects will be enrolled in the study. A software of big data will be used to do a sub study for comparing the results obtained through this software tool against results obtained through Gold standard classical methods used in this prospective observational study (the descriptive assessment of severe asthma prevalence and the prospective evolution of subjects).

ELIGIBILITY:
Inclusion Criteria

* Group A: Subjects with Severe asthma can be enrolled, when they fulfill the following criteria:
* Subjects >= 18 years
* Subjects diagnosed with "severe asthma" defined as asthma that requires high-dose inhaled corticosteroids (ICS) plus Long-Acting Beta2-Agonist (LABA), leukotriene modifier/ theophylline in the last 12 months or continuous/almost continuous treatment with systemic glucocorticosteroids (CS) for >= 50% of the previous year to maintain control of asthma
* Subjects treated with ICS/LABA, with the maximum dose recommended by Specific Product Characteristics (SPC).
* Subjects who give voluntary written informed consent after explanation of study´s procedures.
* Group B: Subjects with Non-Severe asthma can be enrolled, when they fulfill the following criteria:
* Subjects >= 18 years
* Subjects diagnosed with non-severe asthma per GINA Guidelines Classification
* Subjects who give voluntary written informed consent after explanation of study´s procedures

Exclusion Criteria

* Subjects who are not able to complete all the follow-ups of the study with all the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The severe asthmatic subjects according to the ATS/ERS Guidelines will enter into the prospective phase of the study. Non-severe asthmatic subjects will be also enrolled as a control group.
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of severe asthmatic subjects at Spanish sites | Up to 12 months
  Assessment will be done based on the type of hospital, department type of hospital or clinic, sources of the service and number of asthmatic subjects diagnosed according to GEMA guidelines.

SECONDARY OUTCOMES:
Number of subjects with sociodemographic characteristics of severe asthmatic subjects compared to non-severe asthmatic subjects | Up to 12 months
  Subjects with different age, gender, ethnicity, education, occupational status, marital status, physical examination, smoking status, family history, co-morbidities and allergies will be compared for descriptive analysis of sociodemographic characteristics of subjects with severe asthma and non-severe asthma participating in this study.
Number of subjects with clinical characteristics of severe asthmatic subjects compared to non-severe asthmatic subjects | Up to 12 months
  Subjects with asthma severity, age of asthma onset, laboratory tests, biomarkers, skin prick test, airflow tests, asthma symptoms and exacerbations will be compared for clinical characteristics analysis of subjects with severe asthma and non-severe asthma participating in this study.
To estimate the prevalence of different phenotypes in severe asthma | Up to 12 months
  Prevalence of different severe asthma phenotypes (allergic, base on prick test, Immunoglobulin E (IgE), eosinophilic, based on eosinophils counts >= 300 cells/millimeter cubed in blood samples in the previous year, obesity, based on the absence of positive prick test, IgE or high eosinophils counts in blood sample; neutrophilic, just in case eosinophils in sputum are available.
Number of subjects who comply with eligibility criteria to receive biological treatment for severe asthma | Up to 12 months
  Number of exacerbations; Oral Corticosteroid (OCS) treatment; Number of visits to emergency room (ER) and/or hospitalization within the last 12 months, sputum eosinophils (if done), eosinophils in blood, IgE (specific and total), forced expiratory volume-one second (FEV1), Asthma Control Test (ACT), percentage of reversibility will be assessed.
Number of subjects evolved with severe asthma and non-severe asthma at 6 and 12 months from baseline | Up to 12 months
  Exacerbations; visits to emergency room; changes in treatment or dose increase, add-on therapy addition, Disease control (3-score change in ACT), Disease control state (uncontrolled, partially controlled, well controlled) according to guidelines, Quality of life (4-score change in SGRQ), mortality will be assessed.
Number of subjects evolved with severe asthma in comparison with non severe asthma at 6 and 12 months | Up to 12 months
  Subjects with severe and non severe asthma at 6 and 12 months will be compared.
To assess the social impact of subjects with severe asthma in comparison with non-severe asthmatic subjects in terms of Health Related Quality of Life (HRQoL) | Up to 12 months
  Health Related Quality of Life (HRQoL) will be analyzed from the SGRQ Questionnaire scores. Scores will be expressed as percentage of overall impairment, where 100 represents worst possible health and 0 indicates best possible health status.
To assess the use of healthcare resources (direct and indirect) in subjects with severe asthma and non-severe asthma | Up to 12 months
  Direct resources will include number of inpatient admissions, emergency and hospitalized visits, tests to be conducted, etc. on patients with severe asthma. The medical resources used (tests, admissions, etc.) will be analyzed descriptively during the observation period. The direct cost will be calculated by taking into account the resources used and unit costs at a local level. Indirect resources will include reduced productivity of patients with severe asthma through an ad-hoc questions like total number of work days lost due to asthma in the last 6 months.
To predict evolution of subjects with severe and non-severe asthma at month 6 and month 12, based on the physician's experience and knowledge, compared to results obtained through monitoring | Up to 12 months
  The variables to be predicted will be exacerbations; visits to ER; changes in treatment or dose increase; add-on therapy addition; disease control (3-score change in ACT); disease control state (uncontrolled, partially controlled, well controlled) according to guidelines, Quality of life (4-score change in SGRQ) and mortality will be assessed.
To establish the determinant factors clinicians use, to predict subjects evolution | Up to 12 months
  FEV1 (pre & post), percentage reversibility FEV1, number of exacerbations, use of rescue medication, changes to the treatment required, need for adding a biological treatment, concomitant diseases or comorbidities, asthma symptoms; tobacco, eosinophils in blood or sputum, Asthma Control measured by ACT, number or hospitalizations; number of emergency department visits; dose of inhaled glucocorticosteroids, need and dose of oral glucocortocosteroids, mortality, adherence to medication, inhaler technique, fractionated exhaled nitric oxide level (FeNO), Body Mass Index (BMI), GINA treatment Step, living in a rural environment, chronic obstructive pulmonary disease (COPD), male sex, black race, lower educational level will be the determining factor for clinicians.
To test if the calculated prevalence using a specific software is similar to the prevalence of severe asthma obtained through monitoring using gold standard | Up to 12 months
  This will provide a descriptive comparison between the gold standard data and the software's prediction.
To compare the prediction in the evolution of subjects with severe asthma at 6 and 12 months, based on the aggregated information collected in the last 5 years previous to the start of the observational study with the prediction done by the physician | Up to 12 months
  This will provide a descriptive comparison between the clinician's prediction and the software's prediction.
To compare the software's prediction in the evolution of subjects with severe asthma at 6 and 12 months with the results obtained by monitoring in the observational study | Up to 12 months
  Gold standard data collected by monitoring will be compared against the real data.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Spain (25):
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Elda (Alicante)
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Loja/ Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Murcia (El Palmar)
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valdemoro/Madrid
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Xátiva-Valencia
  - GSK Investigational Site, Zaragoza

REFERENCES:
- [Background] Almonacid Sanchez C, Melero Moreno C, Quirce Gancedo S, Sanchez-Herrero MG, Alvarez Gutierrez FJ, Banas Conejero D, Cardona V, Soriano JB. PAGE Study: Summary of a Study Protocol to Estimate the Prevalence of Severe Asthma in Spain Using Big Data Methods. J Investig Allergol Clin Immunol. 2021 Jul 26;31(4):308-315. doi: 10.18176/jiaci.0483. Epub 2020 Jan 23. PMID 31983679